CLINICAL TRIAL: NCT05908071
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Study to Evaluate the Efficacy and Safety of SHEN26 Capsule in Adult Participants With Mild to Moderate COVID-19
Brief Title: Study Evaluating SHEN26 Capsule in Patients With Mild to Moderate COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Kexing Pharmaceutical Co., Ltd. (Network)
Responsible Party: Sponsor
Organization: Kexing Biopharm Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KXZY-SHEN26-301
Record Dates: First submitted 2023-06-15; First posted 2023-06-18 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHEN26 (Experimental): Participants will receive SHEN26 400mg twice daily for 5 days.
  Interventions: Drug: SHEN26 capsule
- SHEN26 placebo (Placebo Comparator): Participants will receive SHEN26 placebo twice daily for 5 days.
  Interventions: Drug: SHEN26 placebo

INTERVENTIONS:
Drug: SHEN26 capsule — Capsule administered orally after meals.
  Arms: SHEN26
Drug: SHEN26 placebo — Capsule administered orally after meals.
  Arms: SHEN26 placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-parallel-controlled phase III clinical trial. It is designed to evaluate the efficacy and safety of SHEN26 capsules in Chinese adult patients with mild to moderate COVID-19

ELIGIBILITY:
Inclusion Criteria:

1. Participants ≥18 years of age, male or female.
2. The subjects were classified as mild or moderate COVID-19, confirmed SARS-CoV-2 infection 72 hours prior to randomization.
3. Initial onset 2 of 11 COVID-19 symptoms within 72 hours before randomization, respiratory and feverish symptoms must be included.
4. Female subjects of childbearing age must have a negative urine pregnancy test during the screening.Fertile participants must agree to take effective contraceptive measures.
5. Understand the procedures and methods of this clinical trial, after fully informed and they participate voluntarily and sign the informed consent form.

Exclusion Criteria:

1. Known hypersensitivity to any ingredient in the experimental drug.
2. Patients with severe or critical COVID-19.
3. With abnormal liver function observed at the time of screening: total bilirubin ≥ 2 × upper limit of normal (ULN), or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 3 × ULN.
4. Subjects with liver diseases, including but not limited to the following diseases, which may affect the safety or efficacy evaluation of subjects during the trial as assessed by the investigator:primary biliary cirrhosis、Child-Pugh Class B or C、acute liver failure.
5. Subjects with known human immunodeficiency virus (HIV) infection.
6. Abnormal renal function observed at the time of screening: serum creatinine ≥ 1.5×ULN;or patients receiving continuous renal replacement therapy, hemodialysis, and peritoneal dialysis at the time of screening.
7. Subjects with acute exacerbation of chronic respiratory diseases.
8. Suspected or confirmed acute systemic infections other than COVID-19 observed at the time of screening.
9. Complications requiring surgery before randomized trial or during the entire trial period and major surgery operated 14 days before the randomized trial,or life-threatening comorbidities considered by the investigator within 30 days before the randomized trial.
10. Cardiovascular diseases meeting any of the following criteria:History of myocardial infarction within the past 12 months、Unstable angina、Clinically significant and uncontrollable cardiac arrhythmias、History of stroke or transient ischemic attack requiring drug treatment in the past 12 months、Congestive heart failure of grade ≥ II assessed by New York Heart Association (NYHA)、Localized edema of grade ≥3、Clinically uncontrolled hypertension.
11. Received SARS-CoV-2 monoclonal antibody treatment or prevention within 30 days before the randomized trial.
12. Received convalescent COVID-19 patient plasma or COVID-19 human immunoglobulin therapy within 30 days before the randomized trial.
13. Have taken antiviral drugs within 30 days before the randomized trial.
14. Have taken any COVID-19 vaccine within 3 months or have been infected with new coronavirus within 3 months before the randomized trial.
15. Pregnant and lactating women.
16. Have participated in other clinical trials or are using experimental drugs within 3 months before the randomized trial.
17. Under other conditions that are not suitable for participating in this trial assessed by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2023-05-13 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Time to 11 COVID-19 Symptom Resolution by Day 28 | Day 1 up to 28
  The time from the start of treatment to the time when 11 COVID-19 symptoms get scores of 0 for two consecutive days

SECONDARY OUTCOMES:
Change of viral load compared to the baseline | Baseline, Day 3, and Day 5
Time to 5 COVID-19 Symptom Resolution by Day 28 | Day 1 up to 28
  The time from the start of treatment to the time when 5 COVID-19 symptoms get scores of 0 for two consecutive days
Change of viral load compared to the baseline | Baseline, Day 7
Proportion of participants who are negative for SARS-CoV-2 nucleic acid test | baseline, Day 3, Day 5, and Day 7
Time to sustained alleviation of 11 COVID-19 symptoms | Day 1 up to 28
  The time from the start of treatment to the time when 11 COVID-19 symptoms get scores of 0 or 1 for two consecutive days
Proportion of Participants with COVID-19 related Hospitalization | Day 1 up to 28
Proportion of severe or critical Participants | Day 1 up to 28
Proportion of Participants with All-cause Death | Day 1 up to 28
AE | Day 1 up to 28
  Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital Of Guangzhou Medical University, Guangzhou, Guangdong, China